CLINICAL TRIAL: NCT05709392
Title: Preterm DElayed Cord Clamping and Early Skin-to-Skin Contact
Brief Title: Preterm DElayed Cord Clamping and Early Skin-to-Skin Contact: PreDECESS
Acronym: PreDECESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Thomas Abrahamsson, MD, PhD, Associate Professor, Ostergotland County Council, Sweden
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PreDECESS
Record Dates: First submitted 2022-12-12; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Bonding; Stress; Breastfeeding; Child Development; Adverse Events
Keywords: adverse events
MeSH Terms: conditions — Breast Feeding | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Comparison of a cohort of premature infants born in gestational week 30+0 till 34+6 taken care of at birth in the traditional way and another cohort of infants taken care of with a new method. The study will be prospective and the control group will be enrolled first before and the active group after the new method has been introduced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Delayed cord clamping and early skin-to-skin contact — A new method for taking care of remature infants born in gestational weeks 30+0-34+6 will be introduced with delayed cord clamping and early skin-to-skin-contact with a parent. If the infant needs help with the breathing this can be given during the time when the cord is still intact.

SUMMARY:
The PreDECESS trial is a prospective study where that will evaluate a new method taking care of premature infants in gestational weeks 30+0 to 34+6 at birth. The new method includes delayed cord clamping and early skin-to-skin contact with a parent. Two populations of infants with their parents will be compared. Infants taken care of in the traditional way before the new method is introduced, and infants taken care of with the new method when it is being introduced.

Primary question:

Does delayed cord clamping and early skin-to skin contact (SSC) lead to better bonding between parents and their infants?

Secondary questions:

Are there any potential adverse effects with delayed cord clamping and early skin-to skin contact (SSC)? Is there a difference in infants level of bilirubin, haemoglobin or proBNP? Is there a difference in infants growth? Is there a difference in infants neurological development? Is there a difference in infants and parents level of stress? Is there a difference in mothers production of breastmilk, frequency of breastfeeding or experience of breastfeeding? Is there a difference in parents mood? How do parents of preterm infants experience giving birth of their preterm baby before and after the introduction of the new method?

DETAILED DESCRIPTION:
A new method taking care of premature infants at birth is going to be introduced in several hospitals in Sweden. The new method includes delayed cord clamping (> 3 minutes) and early skin-to-skin contact with a parent. If the infant needs help with the breathing this can be given during the time when the cord is still intact. This method is different from the traditionally way used for the moment when the the cord is clamped soon after the infant is born and bring the infant to a resuscitation table, often outside the delivery room, to stabilize the infant, for example with support for the breathing with ventilation, CPAP (Continuous Positive Airway Pressure) or intubation.

The PreDECESS trial will study how this delayed cord clamping and skin-to-skin contact will affect the infants and their parents.

The study will have a cohort of premature infants taken care of at birth in the traditional way and another cohort of infants taken care of with the new method. The study will be prospective and the control group will be enrolled first and the active group after the new method has been introduced. It will be multi-center study and hospitals in Linköping, Norrköping, Kalmar, Lund and Huddinge will participate. Infants born in gestational weeks 30+0-34+6 through vaginal delivery and admitted to neonatal ward in Sweden will be included.

The trial is going to study bonding with Swedish Mother-to-Infant Bonding Scale (S-MIBS) and Postpartum Bonding Questionnaire (PBQ). Both parents will also fill in questionnaires for evaluation of depression which might have an impact on bonding, Edinburgh Postpartum Depression Scale (EPDS). There might be connections between bonding and breast-feeding and for that analysis we will use Breastfeeding Self efficacy scale (BSES-SF), a questionary which mothers will answer. The infant's neurological development will be evaluated with a questionary to parents, Ages and Stages Questionnaires (ASQ-3). Infants and parents stress will be measured with cortisol and oxytocin in saliva. The infant's temperature, heart frequency, oxygen saturation, oxygen level and need of respiratory assistance for the first three hours after they are born will be documented. Blood sugar, haemoglobin and bilirubin will be taken as part of the clinical practice. ProBNP will be taken when other laboratory parameters are taken as an indicator of heart function. Residual blood in the placenta after cord clamping will be measured. Data from the neonatal period will be collected from the Swedish Quality Register (www.snq.se), and maternal data will be collected from the Swedish Pregnancy Register (www.graviditetsregistret.se).

A validation of the Swedish Mother-to-Infant Bonding Scale (S-MIBS) will be a part of the trial since this has not been done on premature infants.

A qualitative study where we will interview parents to explore their experiences with premature birth, will also be part of the trial. Parents from both epochs, before and after introduction of the new method, will be asked to be included in the sub study. This qualitative part will be done in the hospitals in Linköping and Norrköping.

Cortisol and oxytocin in saliva before and after the introduction of the new method will be analysed as stress markers.

At least 63 infants in the controlgroup has to be included. This makes it possible to analyse two of our most important questions. The first is hypothermia that is a risk factor with the new method. Thermal control has previously been documented as a cornerstone in a study with immediate skin-to skin contact with parents for premature infants born in gestational weeks 28+0 to 31+6. The second important question is the validation of the Swedish Mother-to-Infant Bonding Scale(S-MIBS). After 63 mothers in the controlgroup have answered S-MIBS we will do an interim analysis to decide the final number participants needed in the trial. If the differences are small between the control group in our study and the suspected outcome in the active group (assumed from normal material previously described in a study where S-MIBS were validated on mothers to healthy fullborn infants by our research group), there will be needed very many infants to prove differences between the two groups. Therefore the study has an upper limit set on 6 months as time for inclusion of the control group at every study site. However, the inclusion will continue until at least 126 infants have been included, ie the inclusion time could be longer than 6 months in that situation.

Intention to treat analyses will be applied. Per protocol analyses will also be done including only infants and mothers in each study group that have followed the study protocol. In the control group mothers should not have skin-to-skin contact with the infants for more than 5 minutes during the first 10 minutes and more than 30 minutes for the first 2 hours to participate in the per protocol analysis. The same applies to the infants, but for some safety analyses there must also not have been delayed cord clamping (> 3 minutes). In the interventiongroup mothers and/or partners should have skin-to-skin contact with the infant all the time except when procedures like resuscitation or insertion of an intravenous line has to be done. The infant should have delayed cord clamping according to the criteria. Sensitivity tests of intention to treat analyses can be done with help from the per protocol analyses.

Descriptive statistics will be used for all quantitative outcome measures: mean ± standard deviation and median ± interquartile range. For qualitative outcome measures proportions and/either percent will be used.

For both primary and secondary outcomes Chi2 test (or Fisher´s exact test if any suspected value is less than 5 )will be used to calculate dichotomous values, t-test to calculate continous data which are normally distributed and Mann-Whitney U test for not normally distributed data. For correlation analysis Pearson and Spearman will be used. Regression models (multiple linear, Cox proportional hazards depending on sort of data) will be used to adjust for potential confounders like gestational week, birth wight, gender, APGAR-score and study site. Relative effect of the intervention will be describes with 95% confidence intervals. All analysis will be given account with two-sides 5 % level of significance.

Approval by the Swedish Ethical Review Authority have been obtained for the trial (Dnr 2022-01611-01).

ELIGIBILITY:
Inclusion Criteria:

Infants born in gestational weeks 30+0-34+6 through vaginal delivery and admitted to neonatal ward in Sweden.

Parents must be able to read Swedish.

Exclusion Criteria:

Infants with known disease when an expanded blood volume is expected will be excluded as early cord clamping is recommended (severe anemia, cardiac disease etc).

Infants with known malformations. Infants with severe or moderate asphyxia (defined as APGAR < 4 at 5 minutes of age).

Infants where the physician in charge find it inappropriate with delayed cord clamping.

No time for cord clamping has been registered.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Bonding | Parents will answer the questionnaires 1 week after delivery.
  Bonding will be assessed with a self administrative instrument, Mother-to-Infant Bonding, Scale (S-MIBS), to parents. It consists of eight adjectives, each describing an emotion and parents will answer how well the adjectives correlated to how they felt for the last 7 days on a four-point scale ranging from 0 to 3. The maximum score is 24, with higher values indicating more bonding challenges.
Bonding | Parents will answer the questionnaires 1 week after delivery.
  Bonding will be assessed with a self administrative instrument, Postpartum Bonding Questionnaire (PBQ), to parents. ]. It consists of 25 statements about parents feelings, where parents answer how well statement applies to them on a six-point scales ranging from 0 to 5, with higher values indicating more problems.
Bonding | Parents will answer the questionnaires 1 month after delivery.
  Bonding will be assessed with a self administrative instrument, Mother-to-Infant Bonding Scale (S-MIBS), to parents. It consists of eight adjectives, each describing an emotion and parents will answer how well the adjectives correlated to how they felt for the last 7 days on a four-point scale ranging from 0 to 3. The maximum score is 24, with higher values indicating more bonding challenges.
Bonding | Parents will answer the questionnaires 1 month after delivery.
  Bonding will be assessed with a self administrative instrument, Postpartum Bonding Questionnaire (PBQ), to parents. It consist of 25 statements about parents feelings, where parents answer how well statement applies to them on a six-point scales ranging from 0 to 5, with higher values indicating more problems.
Bonding | Parents will answer the questionnaires when the infants are 2 months old corrected age.
  Bonding will be assessed with a self administrative instrument, Mother-to-Infant Bonding Scale (S-MIBS), to parents. It consists of eight adjectives, each describing an emotion and parents will answer how well the adjectives correlated to how they felt for the last 7 days on a four-point scale ranging from 0 to 3. The maximum score is 24, with higher values indicating more bonding challenges.
Bonding | Parents will answer the questionnaires when the infants are 2 months old corrected age.
  Bonding will be assessed with a self administrative instrument, Postpartum Bonding Questionnaire (PBQ), to parents. It consists of 25 statements about parents feelings, where parents answer how well statement applies to them on a six-point scales ranging from 0 to 5, with higher values indicating more problems.
Bonding | Parents will answer the questionnaires when the infants are 6 months old corrected age.
  Bonding will be assessed with self a administrative instrument, Mother-to-Infant Bonding Scale (S-MIBS), to parents.It consists of eight adjectives, each describing an emotion and parents will answer how well the adjectives correlated to how they felt for the last 7 days on a four-point scale ranging from 0 to 3. The maximum score is 24, with higher values indicating more bonding challenges.
Bonding | Parents will answer the questionnaires when the infants are 6 months old corrected age.
  Bonding will be assessed with self a administrative instrument, Postpartum Bonding Questionnaire (PBQ), to parents. It consists of 25 statements about parents feelings, where parents answer how well statement applies to them on a six-point scales ranging from 0 to 5, with higher values indicating more problems.

SECONDARY OUTCOMES:
Cortisol in saliva | The saliva tests will be done when the infants are 7 ± 1 days, and 1 month corrected age.
  Cortisol in saliva will be taken on infants before and after diaper change. Cortisol in saliva is measured on both parents at the same time.
Oxytocin in saliva | The oxytocin tests will be taken when the infants are 8 ± 1 days old.
  Oxytocin in saliva will be taken on infants and their mothers before, during and after skin-to-skin holding.
Depression in parents | Parents will answer the questionnaire 1 week and 1 month after delivery and when the infants are 2 and 6 months old corrected age.
  Depression will be assessed with a self administrative instrument, Edinburgh Postnatal Depression Scale (EPDS), to parents. It consists of 10 questions rated on a scale ranging from 0 to 3, with higher values indicating more symptoms.
Experience of breastfeeding | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age.
  Mothers experiences of breastfeeding will be evaluated with a self administrative instrument, Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), to mothers. It assess breast-feeding confidence and consists of 33 items scored on a 5-point scale ranging from 1 (not at all confident) to 5 (always confident). As such, total scores can range from 33 to 165, with higher scores reflecting greater levels of breastfeeding self-efficacy.
Breastmilk production | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age. Data from the Swedish Quality Register will be collected after all the infants have been included in the study.
  Mothers breastmilk production will be assessed with an extra question on the questionnaire Breastfeeding Self-Efficacy Scale-Short Form where the mothers will answer what kind of food their infants are eating, mothers own breastmilk or formula, and approximately how big part of each. Data will also be taken from the Swedish Quality Register where it will be registered what kind of food the infants are eating when they are discharged from hospital.
Frequency of breastfeeding | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age. Data from the Swedish Quality Register will be collected after all the infants have been included in the study.
  Mothers frequency of breastfeeding will be assessed with an extra question on the questionnaire Breastfeeding Self-Efficacy Scale-Short Form where the mothers will answer if they are breastfeeding their babies, totally or partly and if party approximately how much. Data will also be taken from the Swedish Quality Register where it will be registered if mothers are breastfeeding when the infants are discharged from hospital, totally or partly.
Childrens growth in weight | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age. Data from the Swedish Quality Register will be collected after all the infants have been included in the study.
  How the children grows will be assessed with an extra question on the questionnaire Breastfeeding Self-Efficacy Scale-Short Form where mothers will answer what the infants weight, length and head circumference was at their latest visit at BVC. Data will also be taken from the Swedish Quality Register where the infants weight, length and circumference at discharge fron hospital will be registered.
Childrens growth in length | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age. Data from the Swedish Quality Register will be collected after all the infants have been included in the study.
  How the children grows will be assessed with an extra question on the questionnaire Breastfeeding Self-Efficacy Scale-Short Form where mothers will answer what the infants weight, length and head circumference was at their latest visit at BVC. Data will also be taken from the Swedish Quality Register where the infants weight, length and circumference at discharge fron hospital will be registered.
Childrens growth in head circumference | Mothers will answer the questionnaire when the infants are 2 and 6 months old corrected age. Data from the Swedish Quality Register will be collected after all the infants have been included in the study.
  How the children grows will be assessed with an extra question on the questionnaire Breastfeeding Self-Efficacy Scale-Short Form where mothers will answer what the infants weight, length and head circumference was at their latest visit at BVC. Data will also be taken from the Swedish Quality Register where the infants weight, length and circumference at discharge fron hospital will be registered.
Childrens neurological development | Parents will answer the questionnaires when the infants are 12 and 48 months old corrected age.
  Neurological development will be assessed with a self administrative instrument, Ages and Stages Questionnaires (ASQ-3) to parents. It is a developmental screening tool that pinpoints developmental progress in children. It covers five areas of child development that includes: communication, gross motor, fine motor, problem solving, personal-social. There are scores for each area: Yes = 10 points, sometimes = 5 points, not yet = 0 points. Total scores are calculated and higher scores indicate more positive outcomes.
Residual blood in placenta | Residual blood will be measured directly after each delivery and registered on a documentation sheet. This will be done with all vaginal deliveries as long as the study is going on.
  Residual amount of blood in placenta after cord clamping will be measured by allowing the blood that is left after the placenta transfusion flow passively out i a bowl.
Temperature | The temperature will be registered on a documental sheet when the infants are 20, 60, 120 and 180 minutes old. This will be done with all vaginal deliveries as long as the study is going on.
  Infants temperature will be measured regularly during the first 3 hours after delivery. Number of infants with temperature < 36,5 will be documented in the report.
Heart frequency, | The heart frequency will be registered on a documental sheet when the infants are 10, 20, 30, 60, 90, 120, 150 and 180 minutes old. This will be done with all vaginal deliveries as long as the study is going on.
  Infants heart frequency will be measured regularly during the first 3 hours after delivery.
Respiratory frequency | The respiratory frequency will be registered on a documental sheet when the infants are 10, 20, 30, 60, 90, 120, 150 and 180 minutes old. This will be done with all vaginal deliveries as long as the study is going on.
  Infants respiratory frequency will be measured regularly during the first 3 hours after delivery.
Oxygen saturation | Oxygen saturation will be registered on a documental sheet when the infants are 10, 20, 30, 60, 90, 120, 150 and 180 minutes old.This will be done with all vaginal deliveries as long as the study is going on.
  Infants oxygen saturation will be measured regularly during the first 3 hours after delivery. Saturation in percent between 0 and 100 will be registered. Number of infants with saturation < 90 percent will be documented in the report.
Respiratory support | Possible need and what kind of respiratory support will be registered on a documental sheet for the first 3 hours after delivery. This will be done with all vaginal deliveries as long as the study is going on.
  Infants need of respiratory support during the first 3 hour after delivery.
Oxygen level | Possible need of extra oxygen will be registered on a documental sheet for the first 3 hours after delivery.This will be done with all vaginal deliveries as long as the study is going on.
  Infants need of extra oxygen during the first 3 hour after delivery. Fraction of inspired Oxygen (FiO2) will be registered.
Ventilation | Possible need of ventilation will be registered on a documental sheet in the delivery room until discharge from the hospital, up to 1 month corrected age. This will be done with all vaginal deliveries as long as the study is going on.
  Infants need of ventilation in the delivery room.
Blood sugar | Tests will be taken as part of the clinical routine and registered on the same documental sheet as all other outcomes described above until discharge from the hospital, up to 1 month corrected age.
  Infants blood sugar will be measured as part of the clinical routine. Hypoglycemia is defined as blood sugar < 2,6.
Bilirubin | Tests will be taken as part of the clinical routine and registered on the same documental sheet as all other outcomes described above until discharge from the hospital, up to 1 month corrected age.
  Bilirubin level will be measured on the skin or in the blood as part of the clinical routine.
Haemoglobin | Tests will be taken as part of the clinical routine and registered on the same documental sheet as all other outcomes described until discharge from the hospital, up to 1 month corrected age.
  Blood haemoglobin level will be measured as part of the clinical routine.
ProBNP | ProBNP will be taken at the same time as PKU, when the infants are between 48 and 72 hours old. This will be done with all vaginal deliveries as long as the study is going on.
  ProBNP in blood will be measured to assess heart function. The test will be taken as part of the clinical routine at the same time as the PKU test which is taken on all babies in Sweden.
Necrotising enterocolitis, NEC | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnosed clinical, radiological or with autopsy. Incidens in both study groups will be reported.
Spontaneous intestinal perforation, SIP | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Focal intestinal perforation. Diagnosed with operation or autopsy. Incidens in both study groups will be reported.
Surgery | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Extensive surgery in the abdomen, thorax or head. Surgery that is reported according to clinical routines in the Swedish Quality Register. Incidens in both study groups will be reported.
Sepsis | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Clinical symptoms och ≥1 positive blood culture and laboratory signs of infection according to the clinical routines. Incidens in both study groups will be reported.
Suspected sepsis | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Clinical symptoms and laboratory signs of infection, but not culture-proven. Incidens in both study groups will be reported.
Pneumonia | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Pathological X-ray confirmed, need of increased respiratory support/oxygen and laboratory inflammatory response.Incidens in both study groups will be reported.
Respiratory distress syndrome, RDS | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  paO2 <6,6 kPa or central cyanosis in air or need of extra oxygen to reach paO2 ≥6.6 and RDS on chest X-ray. Incidens in both study groups will be reported.
Bronchopulmonary dysplasia, BPD | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnose according to clinical routines, usually meaning need of extra oxygen in gestational week 36+0. Incidens in both study groups will be reported.
Interstitial emphysema | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnose on chest X-ray. Incidens in both study groups will be reported.
Pneumothorax | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Pneumothorax, meaning air in the pleural space, that needs to be drained. Incidens in both study groups will be reported.
Neonatal adaption syndrome, NAS | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  The mildest form of respiratory disorder with laboured breathing. Incidens in both study groups will be reported.
Pulmonary adaption disorder, PAS | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  A slightly more pronounced form of respiratory disorder with the same symptoms , but persists longer and with signs of fluid in the lungs on X-ray. Incidens in both study groups will be reported.
Retinopathy of the prematurity, ROP | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnosed by an independent ophthalmologist according to international classification. Incidens in both study groups will be reported.
Intraventricular haemorrhage, IVH | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnosed according to international classification. Incidens in both study groups will be reported.
Periventricular leukomalacia, PVL | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Diagnosed according to international classification. Only cystic periventricular leukomalacia will be registered. Incidens in both study groups will be reported.
Seizures | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Multiple seizures during the first 12 hours. Clinical or on EEG. Incidens in both study groups will be reported.
Persistent ductus arteriosus | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Persistent ductus arteriosus treated with medicine or surgery. Incidens in both study groups will be reported.
Number of days with intensive care | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Need of respirator or CPAP until discharge (not later than gestational week 44+0).
Length of stay at the hospital | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Gestational week and day at discharge (not later than gestational week 44+0).
Mortality | Data will be collected from the Swedish Quality Register after all the infants have been included in the study, approximately between 1 and 8 years from study start.
  Including cause of death. Incidens in both study groups will be reported.
Parents experiences | Parents will be interviewed close to discharge from hospital or when their children are still in neonatal home care, up to 3 months corrected age. This will be as long as the study is going on.
  To explore parents' experiences in relation to birth of their preterm baby when delayed cord clamping and early skin-to-skin contact is practiced parents from both epochs will be interviewed.

CONTACTS AND LOCATIONS:
Locations (1):
- Crown Princess Victoria children´s hopsital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided